CLINICAL TRIAL: NCT05611983
Title: Experience and Feasibility of Methods for Early Sensory Training Phase 1 - From a User Perspective
Brief Title: Experience and Feasibility of Methods for Early Sensory Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Ulrika Wijk, Principal Investigator, Lund University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2021-03519
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Nerve Injury; Peripheral Nerve Injuries
Keywords: periferal nerve injuries; sensory relearning; rehabilitation; imagery; mirror therapy
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcome assessor/investigator are blinded from which intervention given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Observation fo touch (Active Comparator)
  Interventions: Behavioral: sensory relearning
- Observation of pictures (Active Comparator)
  Interventions: Behavioral: sensory relearning
- Imagery of touch (Active Comparator)
  Interventions: Behavioral: sensory relearning
- Mirror therapy (Active Comparator)
  Interventions: Behavioral: sensory relearning

INTERVENTIONS:
Behavioral: sensory relearning — feasibility of early sensory relearning

SUMMARY:
The good effects of using guided plasticity for a rehabilitative purpose in case of nerve damage have been shown, but a problem that has been presented is that some individuals find it difficult to assimilate these effects due to difficulties in carrying out abstract training or due to a lack of motivation. In early sensory training, the plasticity of the brain is used. Methods for early sensory training that have been described are: 1) mental imagery of touch (mental imagery), 2) observation of touch, 3) mirror training, 4) use of images for visualization of touch. The method needs to be developed and refined to be able to offer individual training plans in order to find a motivating and meaningful form of training.

ELIGIBILITY:
Inclusion Criteria:

* >= 50% injury of N. Medianus/ N. Ulnaris or 100% digital nerve injury dig I and/or dig II
* Ålder: ≥ 18 år

Exclusion Criteria:

* Impaired cognitive ability
* Documented psychiatric diagnosis
* Inability to master the Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
PETS - The Problematic Experience of Therapy Scale | 4 weeks post intervention
  questionnaire, 5-grading scale from "strongly agree" to 'strongly disagree'' to all items in a subscale are recoded as ''no barriers'', and all other scores are recoded as ''some barriers or doubts'' for completing the therapy/sensory relearning.
ESRQ - Early sensory relearing questionaire | 4 weeks post intervention
  questionnaire, 5-grading scale from "strongly agree" to 'strongly disagree''

CONTACTS AND LOCATIONS:
Overall Officials: Lars Dahlin, Prof, Study Chair — Lund University/Region Skane
Locations (1):
- Skane university hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vikstrom P, Carlsson I, Rosen B, Bjorkman A. Patients' views on early sensory relearning following nerve repair-a Q-methodology study. J Hand Ther. 2018 Oct-Dec;31(4):443-450. doi: 10.1016/j.jht.2017.07.003. Epub 2017 Sep 28. PMID 28967458
- [Background] Rosen B, Vikstrom P, Turner S, McGrouther DA, Selles RW, Schreuders TA, Bjorkman A. Enhanced early sensory outcome after nerve repair as a result of immediate post-operative re-learning: a randomized controlled trial. J Hand Surg Eur Vol. 2015 Jul;40(6):598-606. doi: 10.1177/1753193414553163. Epub 2014 Oct 7. PMID 25294735
- [Background] Bassolino M, Campanella M, Bove M, Pozzo T, Fadiga L. Training the motor cortex by observing the actions of others during immobilization. Cereb Cortex. 2014 Dec;24(12):3268-76. doi: 10.1093/cercor/bht190. Epub 2013 Jul 29. PMID 23897648
- [Background] Duffau H. Brain plasticity: from pathophysiological mechanisms to therapeutic applications. J Clin Neurosci. 2006 Nov;13(9):885-97. doi: 10.1016/j.jocn.2005.11.045. Epub 2006 Oct 17. PMID 17049865
- [Result] Vikstrom P, Rosen B, Carlsson IK, Bjorkman A. The effect of early relearning on sensory recovery 4 to 9 years after nerve repair: a report of a randomized controlled study. J Hand Surg Eur Vol. 2018 Jul;43(6):626-630. doi: 10.1177/1753193418767024. Epub 2018 Apr 16. PMID 29661095